CLINICAL TRIAL: NCT05744596
Title: Assessment of the Role of INCisura Biopsy in incrEASing the Stage of Chronic Gastritis
Brief Title: Assessment of the Role of Incisura Biopsy in the Staging of Chronic Gastritis
Acronym: INCREASE
Status: Recruiting | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, Andrei Voiosu, Principal investigator, Clinical Hospital Colentina
Other Study IDs: INCREASE
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic; Gastritis, Atrophic
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gastric mucosa biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incisura biopsy +: this arm has the incisura biopsy scored and added in the OLGA final stage
  Interventions: Other: Incisura biopsy analysis
- Incisura biopsy -: this arm only has corpus and antrum biopsies scored for OLGA staging

INTERVENTIONS:
Other: Incisura biopsy analysis — a pathologist blinded to the other biopsies analyzes the biopsy from the incisura
  Groups: Incisura biopsy +

SUMMARY:
This prospective multicenter study investigates the added benefit of incisura biopsy to correct identification of patients with high-risk chronic gastritis (OLGA stages III-IV). It compares a biopsy protocol with and without a single incisura biopsy in a non-inferiority design.

DETAILED DESCRIPTION:
We will perform a prospective, multicenter, randomized controlled trial of 2 different gastric biopsy protocols. Our hypothesis is that a gastric mapping protocol not including the incisura biopsy ("I-": 2 biopsies from the antrum, 2 from the corpus) is non-inferior to the conventional 5-biopsy approach ("I+": 2 biopsies from the antrum, 2 from the corpus, 1 from the incisura). The primary endpoint of this study is to assess the sensitivity of the "I-" protocol in diagnosing high-risk precancerous chronic gastritis (OLGA/OLGIM stages III or IV) compared to the assumed gold standard of histology based on the "I+" protocol.

In designing the study, we opted for a non-inferiority paired design with high-risk chronic gastritis as a primary binary outcome and a non-inferiority margin (Δ) of 5 % (two-sided 95% CI). The non-inferiority margin was established according to clinical judgement, taking into consideration the significance of a missed diagnosis of high-risk preneoplastic condition and previous estimates of the added value offered by the added incisura biopsy. With a power of 80% and a 2-sided α-level set at 0.05, we estimate that 370 subjects are needed to show non-inferiority. Finally, we will enroll 400 subjects to compensate for eventual exclusions or protocol deviations.

Cohen's kappa will be used to rate intra and inter-observer concordance for pathologists.

An intermediary analysis for futility is scheduled after 100 patients (25%) are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* indication to perform upper GI endoscopy for diagnosis or surveillance

Exclusion Criteria:

* lack of informed consent, previously diagnosed advanced gastric cancer, incomplete endoscopy, surgically altered stomach

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years undergoing upper GI endoscopy are considered eligible for this study, regardless of gender, age or indication.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of OLGA III-IV | at time of enrollment
  number of patients with confirmed OLGA III-IV

SECONDARY OUTCOMES:
prevalence of OLGIM III-IV | at time of enrollment
  number of patients with confirmed OLGIM III-IV

CONTACTS AND LOCATIONS:
Locations (1):
- Colentina Clinical Hospital, Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and images from endoscopy and pathology are shared between participating centers according to the protocol.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available during the study period, after enrollment of all participants. Possible usage of the anonymized database will be discussed by study investigators.
Access Criteria: reasonable request